CLINICAL TRIAL: NCT06498115
Title: Effect of Prophylactic Intravenous Norepinephrine Infusion on Maternal Hypotension After Combined Lumbar and Epidural Anaesthesia for Caesarean Section
Brief Title: Norepinephrine on Maternal Hypotension After Combined Lumbar and Epidural Anaesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Third People's Hospital of Bengbu (Other Government)
Responsible Party: Principal Investigator, Chengfei Xu, doctor-in-charge, The Third People's Hospital of Bengbu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-k21
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Maternal Hypotension
Keywords: norepinephrine; maternal hypotension
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Norepinephrine Bolus (Experimental): Participants in this arm will receive norepinephrine as a bolus dose to treat maternal hypotension during cesarean section under spinal anesthesia. The dosage will be determined using the upper and lower sequential distribution method (UDM). The aim is to investigate the effective dose (ED50 and ED95) of norepinephrine in maintaining maternal blood pressure stability and optimizing maternal outcomes during the procedure.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Participants in this arm will receive norepinephrine as a bolus dose to treat maternal hypotension during cesarean section under spinal anesthesia. The dosage will be determined using the upper and lower sequential distribution method (UDM). The aim is to investigate the effective dose (ED50 and ED95) of norepinephrine in maintaining maternal blood pressure stability and optimizing maternal outcomes during the procedure.

SUMMARY:
Norepinephrine has emerged as a potential alternative for stabilizing blood pressure during spinal anesthesia for cesarean section, purportedly maintaining maternal heart rate and cardiac output more effectively than phenylephrine. However, its application as an intravenous bolus for treating hypotension remains underexplored. Consequently, this current investigation aimed to determine the ED50 and ED95 of norepinephrine for managing maternal hypotension during cesarean section. A prospective trial enrolled 100 patients undergoing elective delivery under spinal anesthesia, with norepinephrine dosage determined using the upper and lower sequential distribution method (UDM).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria included women undergoing elective caesarean section undergoing combined lumbar and rigid anaesthesia, healthy singleton pregnancies at full term (more than 37 weeks gestation), American Society of Anaesthesiologists physical status I or II, body weight between 50-100 kg, height between 150-180 cm, and fasting for more than 8 hours.

Exclusion Criteria:

The exclusion criteria included individuals with hypertension, cardiovascular diseases, preeclampsia, arrhythmias, diabetes mellitus, spinal cord malformations, abnormal fetal conditions, and those who declined to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intravenous norepinephrine to maintain maternal systolic blood pressure 80% above baseline before fetal delivery. | From the initiation of anesthesia to the delivery of the fetus.
  Intravenous norepinephrine pumped to maintain maternal systolic blood pressure 80% above its basal value prior to delivery of the foetus

SECONDARY OUTCOMES:
Intraoperative adverse reactions | Perioperative period
  Dizziness, chest tightness, nausea, vomiting, bradycardia, secondary hypertension and other adverse reactions
Number of remedial drugs | Perioperative period
  Includes incidence of remedial use of atropine, incidence of remedial use of norepinephrine.
Neonatal Apgar score | Immediately After delivery of the foetus
  Neonatal 1-min and 5-min Apgar scores

CONTACTS AND LOCATIONS:
Overall Officials: Liang Cheng, Study Director — The Third People's Hospital of Bengbu
Locations (1):
- The Third People's Hospital of Bengbu, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No